CLINICAL TRIAL: NCT01549028
Title: The Prevalence, Correlations and Effectiveness of Intervention of Osteoporosis in COPD Patients
Brief Title: Osteoporosis in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ho Shu-Chuan, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100-2225A3
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: COPD,; Osteoporosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile-based PR program. (Experimental): Home based mobile PR program for 3 months.
  Interventions: Behavioral: mobile-based PR program.

INTERVENTIONS:
Behavioral: mobile-based PR program. — Patients will be trained and monitored by mobile-based pulmonary rehbailitation program. By mobile, patients could undergo exercise training at home and the information of training parameters will be send to investigator. Investigator could monitor these patients by mobile. Patients will return to visit physian and receive six-minutes walking test to measure outcomes 3 months and 1 year later after mobile-based pulmonary rehabilitation program.

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) are at increased risk of osteoporosis and fractures. Osteoporosis, however, may be equally as disabling as COPD, and may impair respiratory function even further if the patient experiences vertebral compressions.

In this study, we will survey the prevalence, correlations and effectiveness of intervention of osteoporosis in COPD patients.

DETAILED DESCRIPTION:
COPD has a multiple etiology and organ impaired inflammatory disease. In clinical characteristic include airway inflammatory response, cili mobility impairment and lung consolidation change; the others change includes: other functional impairments such as malnutrition, body mass loss, osteogenesis and osteoporosis. The prevalence of osteoporosis and osteopenia patients is generally higher than in healthy subjects and some other chronic disease. Patients with chronic obstructive pulmonary disease are at increased risk of osteoporosis and fractures. Risk factors such as smoking, advanced age, physical inactivity, malnutrition, and low weight may be responsible, but a number of pathophysiological explanations including the presence of a chronic inflammatory state with increased levels of proinflammatory cytokines and protein catalytic enzymes may also be involved. The use of oral glucocorticoids is also a significant risk factor. Osteoporosis, however, may be equally as disabling as COPD, and may impair respiratory function even further if the patient experiences vertebral compressions and loss of height The number of patients with osteoporosis is rising and osteoprosis becomes an important medical and public health issue as the population gets older including Taiwan. Osteoporosis is a silent disease and it is thus important to screen for osteoporosis institute treatment an dreduce fracture incidence. In this study, we will survey the prevalence, correlations and effectiveness of intervention of osteoporosis in COPD patients. This study purpose hope can understand patient's osteoporosis status, pulmonary function impairment and exercise intolerance. Then, we may be can prevent the unnecessary of fracture and maintance of bone mineral contains by the pulmonary rehabilitation program training in osteoporosis COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* with chronic obstructive pulmonary disease.
* with osteoporosis.

Exclusion Criteria:

* could not receive six-minutes walking test.
* could not receive mobile-based pulmonary rehabilitation.
* acute exacerbation of COPD recent 3 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
exercise tolerance. | 3 months
  Exercise tolerance will be measured by six-minutes walking test after trainsing with 3 months mobile-based pulmonary rehabilitation program. Wlaking distences will be the primary outcome measurement.

SECONDARY OUTCOMES:
Inflammatory cytokine of patients. | 3 months and 1 year
  Inflammatory cytokine of enrolled patients including IL-6、IL-8、TNF-α & CRP before and 3 months, 1 year after moble-based pulomonary rehabilitation program will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chuan Ho, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan

REFERENCES:
- [Background] Liu WT, Huang CD, Wang CH, Lee KY, Lin SM, Kuo HP. A mobile telephone-based interactive self-care system improves asthma control. Eur Respir J. 2011 Feb;37(2):310-7. doi: 10.1183/09031936.00000810. Epub 2010 Jun 18. PMID 20562122
- [Background] Liu WT, Wang CH, Lin HC, Lin SM, Lee KY, Lo YL, Hung SH, Chang YM, Chung KF, Kuo HP. Efficacy of a cell phone-based exercise programme for COPD. Eur Respir J. 2008 Sep;32(3):651-9. doi: 10.1183/09031936.00104407. Epub 2008 May 28. PMID 18508824